CLINICAL TRIAL: NCT01032213
Title: Effect of Magnesium Sulphate on Postoperative Coagulation as Measured by Thromboelastography
Brief Title: Effect of Magnesium Sulphate on Coagulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Dr., Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TEG/Mg
Record Dates: First submitted 2009-12-10; First posted 2009-12-15 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Myoma
MeSH Terms: conditions — Myoma | interventions — Magnesium Sulfate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group C (Placebo Comparator): control group
  Interventions: Drug: normal saline
- group M (Experimental): magnesium group
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — Group M received 50 mg/kg of magnesium sulphate on 100 ml of isotonic saline over 10 minutes during the anesthesia induction, followed by the 15 mg/kg/h by continuous infusion during the operation
  Other Names: magnesium sulphate
  Arms: group M
Drug: normal saline — Group S received the same volume of isotonic saline as same method.
  Other Names: isotonic saline
  Arms: group C

SUMMARY:
Arterial and venous thrombotic events are the clinical manifestation of postoperative hypercoagulability. Altered serum magnesium may play a role in the balance of coagulation. In this study, the investigators investigated the effect of magnesium sulphate on the postoperative coagulation change in total intravenous anesthesia (TIVA).

ELIGIBILITY:
Inclusion Criteria:

* ASA Ⅰ-Ⅱ patients undergoing pelviscopic gynecologic operation under general anesthesia.

Exclusion Criteria:

* Pregnancy
* Previous known hematologic disorder
* Recent medication interfering with hemostasis
* Severe anemia
* Liver disease
* Cardiovascular or respiratory disease

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
thromboelastography (TEG) analysis | twice
  1. 10 minutes before the induction of anesthesia
  2. 10 minutes after the recovery from the anesthesia

SECONDARY OUTCOMES:
hemoglobin level | twice
  1. 10 minutes before the induction of anesthesia
  2. 10 minutes after the recovery from the anesthesia
platelet count | twice
  1. 10 minutes before the induction of anesthesia
  2. 10 minutes after the recovery from the anesthesia
international normalized ratio of prothrombin time (INR-PT) | twice
  1. 10 minutes before the induction of anesthesia
  2. 10 minutes after the recovery from the anesthesia
activated partial thromboplastin time (aPTT) | tiwce
  1. 10 minutes before the induction of anesthesia
  2. 10 minutes after the recovery from the anesthesia
serum magnesium level | twice
  1. 10 minutes before the induction of anesthesia
  2. 10 minutes after the recovery from the anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea